CLINICAL TRIAL: NCT06034197
Title: Pilot Open Label Study to Determine the Safety and Efficacy of Fluorescent Probe, VGT-309, to Identify Cancerous Colorectal Lesions During White-Light and Fluorescence Augmented Colonoscopy
Brief Title: Fluorescent Probe VGT-309 to ID Cancerous Colorectal Lesions During Augmented Colonoscopy
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: We are awaiting new stock of the investigational drug.
Sponsor: Stephan Rogalla (Other)
Responsible Party: Sponsor-Investigator, Stephan Rogalla, Clinical Assistant Professor, Medicine - Gastroenterology & Hepatology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-68096; NCI-2024-01204 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VGT-309 (Experimental): Subjects will receive an IV infusion of 0.32 mg/kg VGT-309 12 to 36 hours before a standard of care endoscopy procedure.
  Interventions: Drug: VGT-309

INTERVENTIONS:
Drug: VGT-309 — 0.32mg/kg IV of VGT-309 given 12-36 hours before surgery

SUMMARY:
The purpose of this study is to determine the safety and feasibility of VGT-309 for the visualization of colorectal tumors in real-time using near-infrared (NIR) fluorescence endoscopy. In addition, signatures of 50+ biomarkers will be evaluated in biopsies using CODEX multi-plexing.

ELIGIBILITY:
Inclusion Criteria

1. Adult patients with histologically confirmed distal colorectal adenocarcinoma of any stage.
2. Be willing and able to sign the informed consent and comply with study procedures.
3. Are scheduled to undergo a SOC colonoscopy for restaging following radiochemotherapy or are scheduled to receive a SOC colonoscopy in the OR prior to resection
4. Have acceptable kidney and liver functions at study entry as evidenced by:

   1. ALT/AST < 1.5 times the upper limit of normal,
   2. Creatinine clearance (according to Cockcroft-Gault Equation) > 50 mL/min
   3. Total bilirubin < 1.5 times the upper limit of normal
5. Have an ECOG score of 0-2.
6. Be at least 18 years of age.
7. Female participants must be of non-childbearing potential, or, if of childbearing potential be non-pregnant or lactating and agree to use highly effective contraception from screening through 30 days after probe infusion
8. Male participants, if not surgically sterilized, and if engaging in sexual intercourse with a female partner of childbearing potential, must be willing to use highly effective contraception from screening through 30 days post-dose and agree not to donate semen during this waiting period.
9. Highly effective contraception involves the use of a condom for the male, plus one of the following for the female:

   1. Oral, injectable, implantable, intravaginal, or transdermal hormonal contraceptives, or
   2. Intrauterine device or intrauterine hormone-releasing system. NOTE: Participants who abstain from heterosexual intercourse as their usual and preferred lifestyle, will not be required to use contraception as described above. They are required to maintain abstinence from screening through Day 30, AND Participants in a same sex relationship, must use a barrier form of contraception (e.g., condom, diaphragm) to protect against the transfer of the study drug in any bodily fluids.

Exclusion Criteria:

Inclusion Criteria:

1. Adult patients with histologically confirmed distal colorectal adenocarcinoma of any stage.
2. Be willing and able to sign the informed consent and comply with study procedures.
3. Are scheduled to undergo a SOC colonoscopy for restaging following radiochemotherapy or are scheduled to receive a SOC colonoscopy in the OR prior to resection
4. Have acceptable kidney and liver functions at study entry as evidenced by:

   1. ALT/AST < 1.5 times the upper limit of normal,
   2. Creatinine clearance (according to Cockcroft-Gault Equation) > 50 mL/min
   3. Total bilirubin < 1.5 times the upper limit of normal
5. Have an ECOG score of 0-2.
6. Be at least 18 years of age.
7. Female participants must be of non-childbearing potential, or, if of childbearing potential be non-pregnant or lactating and agree to use highly effective contraception from screening through 30 days after probe infusion
8. Male participants, if not surgically sterilized, and if engaging in sexual intercourse with a female partner of childbearing potential, must be willing to use highly effective contraception from screening through 30 days post-dose and agree not to donate semen during this waiting period.
9. Highly effective contraception involves the use of a condom for the male, plus one of the following for the female:

   1. Oral, injectable, implantable, intravaginal, or transdermal hormonal contraceptives, or
   2. Intrauterine device or intrauterine hormone-releasing system. NOTE: Participants who abstain from heterosexual intercourse as their usual and preferred lifestyle, will not be required to use contraception as described above. They are required to maintain abstinence from screening through Day 30, AND Participants in a same sex relationship, must use a barrier form of contraception (e.g., condom, diaphragm) to protect against the transfer of the study drug in any bodily fluids.

Exclusion Criteria:

1. Pregnant or breastfeeding females
2. They have a known allergy or reaction to ICG, other radiographic contrast agents, or any component of VGT-309.
3. Have congenital long QT syndrome or QTcF > 450ms (males) or >470ms (females) by history or at Screening ECG.
4. They are prisoners, institutionalized individuals, or are unable to consent for themselves.
5. Class 2 or higher obesity, defined by BMI ≥ 35.0.
6. Have any other comorbidity or habit that the Investigator believes will interfere with their ability to comply with and complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety Profile of VGT309 | 18 days
  Safety profile will be measured by assessing number of Grade 2 or higher adverse events which have been determined to be clinically significant and definitely, probably or possibly related.
Feasibility of VGT-309 | 18 days
  Feasibility to visualize colorectal tumors using NIR-endoscopy will be measured by the tumor-to-background ratio (fluorescence intensity of tumor tissue divided by the fluorescence intensity of normal surrounding tissue) and the concordance between white-light endoscopy assessment, histopathological examination and NIR imaging assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Rogalla, M.D., PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States